CLINICAL TRIAL: NCT06415552
Title: Implementation of Online Mindfulness-Based Stress Reduction Tailored for People with Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Simpson (Other)
Responsible Party: Sponsor-Investigator, Robert Simpson, Investigator, Unity Health Toronto
Organization: Unity Health Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Mindfulness for PwMS
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Mindfulness
MeSH Terms: conditions — Multiple Sclerosis | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindfulness-Based Stress Reduction (Other): 8-week Mindfulness-Based Stress Reduction course
  Interventions: Behavioral: Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — Eight iterations of the MBSR course will be delivered, over a total period of 24 months. Each iteration will take place over 8 weeks. Courses would consist of 8 weekly sessions, led by certified mindfulness instructors. Sessions will include core meditation practices, psychoeducation, and home practices.

SUMMARY:
This project aims to implement and investigate a mindfulness-based stress reduction (MBSR) in people with multiple sclerosis (PwMS). The main objective is to implement MBSR intervention for PwMS in a major tertiary care clinic for PwMS. We will iteratively refine the intervention as required based on stakeholder feedback and any other emergent contextual findings.

Participants will be asked to take part in an 8-week MBSR course and report changes in anxiety, depression, quality of life, emotional regulation, self-compassion, mindfulness, and health services use.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years </= 60 years
2. Diagnosis of MS or related condition (Clinically Isolated Syndrome, Neuromyelitis Optica Spectrum Disorder, Chronic Inflammatory Demyelinating Neuropathy)
3. Able to understand spoken and written English
4. Willing to take part in an MBSR course

Exclusion Criteria:

1. Cognitive impairment (<26 on the Montreal Cognitive Assessment)
2. Severe active mental health impairment (psychosis, suicidality)
3. Medical instability (terminal/life threatening inter-current illness)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 24 months
  The investigators will measure the number of participants eligible for and recruited to the study.
Retention | 24 months
  The investigators will measure the percentage of participants who complete outcome data.
Adherence | 24 months
  The investigators will measure the number of participants who completed the mindfulness-based stress reduction course.
Follow-up rates | 24 months
  The investigators will measure the percentage of participants who complete outcome measures pre-intervention, post-intervention, and at 3 months post-intervention.

SECONDARY OUTCOMES:
Quality of Life using the Multiple Sclerosis Impact Scale (MSIS-29) | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Multiple Sclerosis Impact Scale. Items on the scale have a Likert scale from 1-5, with a range of 0-100 total and higher scores indicating greater disability.
Quality of Life using the EuroQol (EQ-5D-5L) | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the EQ-5D-5L. The total score ranges from 1-100, with higher values indicating better perceived health.
Anxiety | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Hospital Anxiety and Depression Scale. The total score ranges from 0-21, with higher values representing increased anxiety symptoms.
Depression | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Hospital Anxiety and Depression Scale. The total score ranges from 0-21, with higher values representing increased anxiety symptoms.
Health services use | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Client Services Receipt Inventory. This instrument is used to collect information on the use of health services.
Emotion regulation | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Difficulties in Emotion Regulation Scale - Short Form. Answers are assessed using a 5-point Likert scale. Higher values indicate greater difficulties in emotion regulation.
Self-compassion | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Self-Compassion Scale - Short Form. The total score ranges from a 1-5 Likert scale, with higher scores representing high self-compassion.
Mindfulness | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Five-facet Mindfulness Questionnaire. Answers are assessed using a 5-point Likert scale. Higher scores in each facet indicate higher levels of mindfulness.
Climate | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Group Climate Questionnaire-Engage Scale. Each item response is measured on a Likert scale from 0-6, with total subscale scores reflecting the average of responses. Higher scores indicate higher group engagement.
Therapeutic alliance | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Working Alliance Inventory. Each item is measured on a 7-point Likert scale, with a range of 36-252 total. Higher scores indicates stronger alliance.
Sleep | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Insomnia Severity Index. The total score ranges from 0-28, with higher scores indicating worse insomnia.
Pain Effects | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Pain Effects Scale. The total score ranges from 6-30, with higher scores indicating greater impact of pain on behavior and mood.
Fatigue | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Modified Fatigue Impact Scale. The total score ranges from 0-84, with higher scores indicating a greater impact of fatigue.
Cognitive function | Measured at baseline, 8-week follow-up, and 3-month follow-up
  Measured using the Symbol Digits Modalities Test. The total score ranges from 0-110, with higher scores indicating better cognitive functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No